CLINICAL TRIAL: NCT00577148
Title: A Double-blind, Randomized, Placebo-controlled, Parallel Group Study of Rimonabant 20 mg Daily for the Treatment of Type 2 Diabetic Patients With Nonalcoholic Steatohepatitis (NASH).
Brief Title: An Efficacy and Safety Study of Rimonabant for Treatment of Nonalcoholic Steatohepatitis (NASH) in Patients With Type 2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision taken in light of demands by certain national health authorities
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC10144; 2007-003013-14 (EudraCT Number)
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Fatty Liver
Keywords: NASH; chronic liver disease
MeSH Terms: conditions — Fatty Liver | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rimonabant (Experimental): Rimonabant 20 mg once daily.
  Interventions: Drug: Rimonabant
- Placebo (Placebo Comparator): Placebo (for Rimonabant) once daily.
  Interventions: Drug: Placebo (for Rimonabant)

INTERVENTIONS:
Drug: Rimonabant — Tablet, oral administration
  Other Names: SR141716; Acomplia
  Arms: Rimonabant
Drug: Placebo (for Rimonabant) — Tablet, oral administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of rimonabant treatment on the histological features of Nonalcoholic Steatohepatitis (NASH) in patients with Type 2 diabetes.

DETAILED DESCRIPTION:
The total duration per patient will be approximately 22 months including a 18-month double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 diabetes mellitus and a diagnosis of NASH

Exclusion Criteria:

* Excessive alcohol use
* Presence of Type 1 diabetes mellitus
* Other chronic liver disease
* Previous or current hepatocellular carcinoma
* Use of medication known to cause steatosis
* Previous bariatric surgery
* Pregnancy or breastfeeding
* Presence of any severe medical or psychological condition that, in the opinion of the investigator, would compromise the patient's safe participation including uncontrolled serious psychiatric illness such a major depression within the last 2 years, and history of other severe psychiatric disorders

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Mean change per year in Non-Alcoholic Fatty Liver Disease [NAFLD] Activity Score (NAS) | Baseline to 18 months

SECONDARY OUTCOMES:
Change from baseline in hepatic fibrosis score | Baseline to 18 months
Change from baseline in serum hyaluronate and hepatic transaminases (AST/ALT) | Baseline to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (24):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Cove, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Shanghai, China
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Zagreb, Croatia
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Makati City, Philippines
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, San Juan, Puerto Rico
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Guildford, Surrey, United Kingdom